CLINICAL TRIAL: NCT02598349
Title: A Phase II Trial of Escalated Dose Proton Radiotherapy With Elective Nodal Irradiation and Concomitant Chemotherapy for Patients With Unresectable, Borderline Resectable or Medically Inoperable Pancreatic Adenocarcinoma
Brief Title: Proton Radiation for Unresectable, Borderline Resectable, or Medically Inoperable Carcinoma of the Pancreas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Proton Collaborative Group (Network)
Collaborators: University of Florida Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAN009-18; UFPTI-1510-PC04 (Other: University of Florida Health Proton Therapy Institute)
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer
Keywords: Unresectable; Borderline resectable
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Proton Therapy; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Proton Radiation with capecitabine (Experimental): The following will be performed in this group: Proton Radiation Therapy with concomitant oral chemotherapy, capecitabine taken on radiation treatment days for 6 weeks. A surgical resection will be performed between 8 and 16 weeks if radiographic studies suggest operability.
  Interventions: Radiation: Proton Radiation; Drug: Capecitabine; Procedure: Surgical resection

INTERVENTIONS:
Radiation: Proton Radiation — Proton Radiation 40.50 Gy relative biological effectiveness (RBE) in 18 fractions to gross disease and elective nodal volume followed by a 22.50 Gy (RBE) in 10 fraction boost to gross disease. Total dose 63 Gy (RBE) in 28 fractions over 6 weeks.
  Other Names: Proton Beam Radiation
Drug: Capecitabine — Concomitant oral chemotherapy, capecitabine 1000mg by mouth twice daily, 5 days a week (M-F) on radiation days only.
  Other Names: Xeloda
Procedure: Surgical resection — Surgery between 8 and 16 weeks of radiotherapy completion if radiographic studies suggest operability.

SUMMARY:
The prognosis for patients with localized pancreatic adenocarcinoma who are not surgical candidates is poor. Patients characterized as having "borderline resectable" disease treated with preoperative chemo-radiotherapy fair somewhat better - although many of these patients are not converted to resectability. It may be argued that intensification of local and regional therapy might 1.) Increase the share of patients able to undergo curative surgery and 2.) Improve the local disease control interval and extend survival for patients who remain unresectable. Therefore, the purpose of this research study is to determine if an increase in the number of surgical resection pancreatic adenocarcinoma is higher than historical data by using a combined treatment of proton radiation with capecitabine (oral chemotherapy).

DETAILED DESCRIPTION:
Participants as part of this research study will receive Proton radiation over 6 weeks with oral chemotherapy (capecitabine) only taken on radiation days.

In addition, If surgery is an option, then surgical resection will be performed at least 8 weeks after treatment with radiation and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven unresectable adenocarcinoma of the pancreas.
* Have either unresectable, borderline resectable or medically inoperable carcinoma of the pancreas, or refusing surgery.
* A biliary obstruction is able to participate as long as a drainage tube is in place prior to starting treatment with Proton radiation,
* Participants of child-producing potential must be willing to use contraception while on treatment and for at least 12 months thereafter.
* Required pretreatment laboratory parameters:

  * Absolute granulocyte count (AGC/ANC) ≥ 1.8 thou/mm3
  * Platelet count ≥ 100,000/mm3
  * Bilirubin < 2 mg/dl
  * ALT/SGPT < 3x upper limit of normal
  * Creatinine < 3 mg/dl

Exclusion Criteria:

* Evidence of distant metastasis.
* Prior surgical resection.
* Previous history of invasive malignancy (except non-melanoma skin cancer and low to intermediate risk prostate cancer) unless the participant has been disease free for 5 years prior to registration.
* Active or untreated infection,
* Pregnant or breastfeeding women or subjects of child producing potential not willing to use medically acceptable contraception while on treatment and for at least 12 months thereafter.
* Previous Radiation to the abdomen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2039-10 (Estimated); Study Completion 2040-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival at 12 months after radiation therapy | Approximately 12 months after radiation therapy.
  The trial is designed to allow detection of an improvement in the 12 month overall survival rate to 75% compared to the expected historical rate of 50%.

SECONDARY OUTCOMES:
Surgical resection rate. | 3 months following the completion of radiation therapy.
  Increase share of marginally resectable and unresectable patients being converted to resectable.

CONTACTS AND LOCATIONS:
Overall Officials: Romaine C. Nichols, MD, Principal Investigator — UF Health Proton Therapy Institute
Locations (4):
- United States (4):
  - University of Florida Proton Therapy Institute, Jacksonville, Florida
  - Northwestern Medicine Chicago Proton Center, Warrenville, Illinois
  - McLaren Proton Therapy Center, Flint, Michigan
  - Inova Schar Cancer Institute, Fairfax, Virginia

REFERENCES:
- [Background] Katz MH, Pisters PW, Evans DB, Sun CC, Lee JE, Fleming JB, Vauthey JN, Abdalla EK, Crane CH, Wolff RA, Varadhachary GR, Hwang RF. Borderline resectable pancreatic cancer: the importance of this emerging stage of disease. J Am Coll Surg. 2008 May;206(5):833-46; discussion 846-8. doi: 10.1016/j.jamcollsurg.2007.12.020. Epub 2008 Mar 17. PMID 18471707
- [Background] Ashman JB, Moss AA, Rule WG, Callister MG, Reddy KS, Mulligan DC, Collins JM, De Petris G, Gunderson LL, Borad M. Preoperative chemoradiation and IOERT for unresectable or borderline resectable pancreas cancer. J Gastrointest Oncol. 2013 Dec;4(4):352-60. doi: 10.3978/j.issn.2078-6891.2013.006. PMID 24294506
- [Background] R. C. Nichols, C. G. Morris, D. Bose, S. J. Hughes, J. A. Stauffer, S. A. Celinski, R. C. Martin II, E. A. Johnson, R. A. Zaiden, M. S. Rutenberg ;O51: Feasibility of pancreatectomy after high dose proton therapy for unresectable pancreatic cancer. (2014) Proceedings to the 1 Annual Meeting for the Particle Therapy Cooperative Group - North America (PTCOG-NA), 27-29 October 2014. International Journal of Particle Therapy: Winter 2014, Vol. 1, No. 3, pp. 759-824.
- [Background] Pawlik TM, Gleisner AL, Cameron JL, Winter JM, Assumpcao L, Lillemoe KD, Wolfgang C, Hruban RH, Schulick RD, Yeo CJ, Choti MA. Prognostic relevance of lymph node ratio following pancreaticoduodenectomy for pancreatic cancer. Surgery. 2007 May;141(5):610-8. doi: 10.1016/j.surg.2006.12.013. Epub 2007 Mar 23. PMID 17462460
- [Background] Winter JM, Brennan MF, Tang LH, D'Angelica MI, Dematteo RP, Fong Y, Klimstra DS, Jarnagin WR, Allen PJ. Survival after resection of pancreatic adenocarcinoma: results from a single institution over three decades. Ann Surg Oncol. 2012 Jan;19(1):169-75. doi: 10.1245/s10434-011-1900-3. Epub 2011 Jul 15. PMID 21761104
- [Background] Lee RY, Nichols RC Jr, Huh SN, Ho MW, Li Z, Zaiden R, Awad ZT, Ahmed B, Hoppe BS. Proton therapy may allow for comprehensive elective nodal coverage for patients receiving neoadjuvant radiotherapy for localized pancreatic head cancers. J Gastrointest Oncol. 2013 Dec;4(4):374-9. doi: 10.3978/j.issn.2078-6891.2013.043. PMID 24294509
- [Background] Dholakia AS, Kumar R, Raman SP, Moore JA, Ellsworth S, McNutt T, Laheru DA, Jaffee E, Cameron JL, Tran PT, Hobbs RF, Wolfgang CL, Herman JM. Mapping patterns of local recurrence after pancreaticoduodenectomy for pancreatic adenocarcinoma: a new approach to adjuvant radiation field design. Int J Radiat Oncol Biol Phys. 2013 Dec 1;87(5):1007-15. doi: 10.1016/j.ijrobp.2013.09.005. PMID 24267969
- [Derived] Rapp CT, Rutenberg MS, Morris CG, Nichols RC. Dose-escalated proton therapy with elective nodal irradiation and concomitant chemotherapy for unresectable, borderline resectable, or medically inoperable pancreatic cancer: a phase II trial. J Gastrointest Oncol. 2022 Jun;13(3):1395-1401. doi: 10.21037/jgo-21-593. PMID 35837200
- See also: Contact the University of Florida Proton Therapy Institute — http://www.floridaproton.org/contact/